CLINICAL TRIAL: NCT05396508
Title: The Effectiveness of Interfacial Injection Applied in Addition to Physical Therapy Applications in Chronic Low Back Pain
Brief Title: Interfacial Injection in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Burcu Metin Ökmen, Assoc.Phd.M.D, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/10-24
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2019-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical therapy (Active Comparator): physical therapy
  Interventions: Procedure: physical therapy
- physical therapy + interfacial injection (Active Comparator): physical therapy + interfascial injection
  Interventions: Procedure: interfacial injection; Procedure: physical therapy

INTERVENTIONS:
Procedure: interfacial injection — 10 ml of bupivacaine and steroid injection was applied between the leaves of the thoracolumbar fascia under the guidance of ultrasonography.
  Arms: physical therapy + interfacial injection
Procedure: physical therapy — protocol including hot pack for 20 min/session, therapeutic continuous Ultrasound (frequency, 1 MHz; intensity 1.5 W/cm2) for 6 min/session, therapeutic exercises for low back muscles. Therapeutic exercises included stretching ,posterior pelvic tilt ,hyperextension ,bridge and cat-camel exercises

SUMMARY:
Its effect on thoracolumbar fascia and low back pain has been investigated in different studies.These studies suggest that the anatomical and histological features of the fascia may have an effect on low back pain. This study aimed to investigate the effectiveness of interfacial injection in patients with chronic back pain.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for more than 6 months;
* Presence of MR findings radiologically diagnosing LDH;
* Numeric rating scale (NRS) > 5

Exclusion Criteria:

* Spinal stenosis;
* Spondylolisthesis;
* Previous lumbar
* Spinal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
NRS | 6 month
  Numeric rating scale(NRS) A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable

SECONDARY OUTCOMES:
ODI | 6 month
  Oswestry Disability Index Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability.The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible
NSAİD | 6 month
  The monthly consumption of NSAIDs was queried (pcs/month)

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, Assoc. PhD., Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa, Turkey (Türkiye)